CLINICAL TRIAL: NCT00362622
Title: Determinants of Compliance With Glaucoma Therapy
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Christopher Girkin, MD, Chairman/Professor, University of Alabama at Birmingham
Other Study IDs: X050826003
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Open Angle Glaucoma
Keywords: Travalert; open angle glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the association between medical, demographic, socioeconomic, and therapeutic differences on compliance with topical glaucoma therapy using the Travalert device.

DETAILED DESCRIPTION:
To determine the association between medical, demographic, socioeconomic, and therapeutic differences on compliance with topical glaucoma therapy using the Travalert device. All participants will have open angle glaucoma.

ELIGIBILITY:
To be eligible to participate in the study, patients had to be (1) 19 years or older; (2) have a diagnosis of open angle glaucoma (OAG) in 1 or both eyes or ocular hypertension; and (3) using a prostaglandin ocular hypotensive medication in 1 or both eyes.

The protocol excluded patients with uncontrolled IOP control, known contraindications to Travoprost, clinically significant systemic disease that would interfere with the study, participation in any other research study within 30 days, or change in systemic medications that may alter IOP within 30 days before recruitment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2005-10; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Girkin, MD, Principal Investigator — University of Alabama at Birmingham; Jason Swanner, MD, Principal Investigator — University of Alabama at Birmingham; Matthew Sapp, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States